CLINICAL TRIAL: NCT05726292
Title: A Randomized Phase II Trial of Neoadjuvant Enzalutamide Plus the Glucocorticoid Receptor Antagonist Relacorilant Versus Placebo for Patients With High-risk Localized Prostate Cancer
Brief Title: A Study of Enzalutamide Plus the Glucocorticoid Receptor Antagonist Relacorilant Versus Placebo for Patients With High-risk Localized Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB22-1318
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma
Keywords: prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — relacorilant; enzalutamide; Sugars; Androgen Antagonists

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: Participants Who Receive Study Drug (Relacorilant) with Hormone Therapy and Enzalutamide (Experimental): All participants in this group will have surgery up to 4 weeks after receiving enzalutamide/relacorilant with hormone therapy. A radical prostatectomy (removal of the prostate and any surrounding tissue that the surgeon thinks may be affected by the cancer).
  Interventions: Drug: Relacorilant; Drug: Enzalutamide; Other: Androgen Deprivation Therapy; Procedure: Radical Prostatectomy
- Group 1: Participants Who Receive Placebo (no study drug) with Hormone Therapy and Enzalutamide (Experimental): All participants in this group will have surgery up to 4 weeks after receiving enzalutamide/placebo (sugar pill in the form of 2 softgel capsules) with hormone therapy. A radical prostatectomy (removal of the prostate and any surrounding tissue that the surgeon thinks may be affected by the cancer).
  Interventions: Drug: Enzalutamide; Other: Placebo (Sugar Pill); Other: Androgen Deprivation Therapy; Procedure: Radical Prostatectomy

INTERVENTIONS:
Drug: Relacorilant — Relacorilant is an antiglucocorticoid which is under development by Corcept Therapeutics for the treatment of Cushing's syndrome. It is being used in this study as an experimental drug combined with other treatments for prostate cancer.
  Arms: Group 1: Participants Who Receive Study Drug (Relacorilant) with Hormone Therapy and Enzalutamide
Drug: Enzalutamide — Enzalutamide, sold under the brand name Xtandi, is a nonsteroidal antiandrogen medication which is used in the treatment of prostate cancer.
  Other Names: Xtandi
Other: Placebo (Sugar Pill) — This would be a sugar pill consisting of 2 softgels. This is not an experimental drug or treatment.
  Arms: Group 1: Participants Who Receive Placebo (no study drug) with Hormone Therapy and Enzalutamide
Other: Androgen Deprivation Therapy — All participants in this study, who meet the requirements to participate, will get Androgen Deprivation Therapy (ADT; a form of hormone therapy) continuously before their radical prostatectomy surgery. As part of this study, ADT consists of one injection every 1-3 months. In this study, ADT is a gonadotropin releasing hormone (GnRH) agonists or antagonist; the choice of which brand of ADT to use is up to your treating physician. GnRH agonists and antagonists are drugs that lower the production of androgens (male hormones) in your body. Prostate cancer cells usually require androgens, such as testosterone, to grow.
  Androgen Deprivation Therapy (ADT) has been approved by United Stated Food and Drug Administration (US FDA) to treat patients with prostate cancer but is not approved to treat patients prior to prostatectomy.
Procedure: Radical Prostatectomy — Radical prostatectomy is surgery to remove the entire prostate gland and surrounding lymph nodes to treat men with localized prostate cancer.

SUMMARY:
Researchers conducting this study hope to learn about the safety and effectiveness of combining two study drugs, relacorilant and enzalutamide, plus androgen deprivation therapy (ADT), also known as hormone therapy. This study is for individuals who have been diagnosed with advanced, high-risk prostate cancer and standard therapies available to treat your disease have not been effective. Participation in this research will last about 3 years and 9 months.

DETAILED DESCRIPTION:
The purpose of this research is to gather information on the safety and effectiveness of combining two study drugs (relacorilant and enzalutamide) with hormone therapy. Doctors leading this study hope to learn if combining these study drugs with hormone therapy is safe and could improve the results of surgery and delay the time to when prostate cancer tumors spread to other parts of the body in individuals with advanced, high-risk prostate cancer who plan to receive a radical prostatectomy (surgical removal of the whole prostate and surrounding tissue).

Prostate cancer cells usually need hormones (called androgens) to grow. One of these hormones is testosterone, which is mostly produced in the testicles. The usual approach for treating prostate cancer after it progresses involves taking medications to decrease or block the development of hormones (including testosterone) so that prostate cancer cells can't continue to grow. This approach is called androgen deprivation therapy (hormone therapy). Enzalutamide is a hormone-blocking medication, which is a standard of care for prostate cancer when it spreads (metastasizes).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed prostatic adenocarcinoma without primary small cell histology
2. Localized disease:

   * Surgical resectability must be documented prior to enrollment
   * No evidence of distant metastatic disease on abdominopelvic imaging, bone imaging

     * Enlarged lymph nodes below the iliac bifurcation (clinical stage N1) is allowed
     * Either cross-sectional abdominopelvic imaging + technetium bone scan or PSMA PET imaging will be acceptable to rule out distant metastatic disease
3. High or very high-risk disease (https://www.nccn.org/professionals/physician_gls/pdf/prostate.pdf) as defined by having one or more of the following:

   * Clinical T3a or higher
   * Histologic Grade Group 4 or 5
   * PSA >20
4. Eastern Cooperative Oncology Group performance status ≤ 1 (Appendix A)
5. Total serum testosterone 100 ng/dL
6. Patients must have normal hepatic function as defined below:

   * Total bilirubin <1.5 X the upper limit of normal (note that in subjects with Gilbert's syndrome, if total bilirubin is >1.5 X ULN, measure direct and indirect bilirubin. If direct bilirubin is ≤1.5 X ULN, the subject may be eligible)
   * AST(SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal
   * Albumin 3.0 g/dL
7. Patients must have normal bone marrow function as defined below:

   * Platelet count (plt) 100,000 /L
   * Hemoglobin (Hgb) 10 g/dL
   * Absolute neutrophil count (ANC) 1500
8. Patients must have adequate renal function as defined below:

   • glomerular filtration rate (GFR) 30 mL/min
9. Ability to understand and the willingness to sign a written informed consent document.
10. Patients with active diabetes mellitus on glucose lowering medications are eligible provided they agree to and are able to self-monitor daily blood glucose levels due to potential risk of lowering glucose levels on relacorilant.
11. Male patient and his female partner who is of childbearing potential must use 2 acceptable methods of birth control (one of which must include a condom as a barrier method of contraception) starting at screening and continuing throughout the study period and for 3 months after final study drug administration. Two acceptable methods of birth control thus include the following:

    * Condom (barrier method of contraception) AND
    * One of the following is required:

      1. Established use of oral, injected or implanted hormonal method of contraception by the female partner;
      2. Placement of an intrauterine device (IUD) or intrauterine system (IUS) by the female partner;
      3. Additional barrier method: Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository by the female partner;
      4. Tubal ligation in the female partner;
      5. Vasectomy or other procedure resulting in infertility (e.g., bilateral orchiectomy), for more than 6 months.

3.2 Exclusion Criteria

1. Therapy with ANY hormonal therapy for prostate cancer (prior 5-alpha-reductase inhibitors for benign prostate disease is allowed but must be discontinued prior to study initiation).
2. Inability to swallow capsules or known gastrointestinal malabsorption.
3. History of other malignancies, with the exception of: adequately treated non-melanoma skin cancer, adequately treated superficial bladder cancer, stage 1 or 2 malignancies that are without evidence of disease, or other cancers curatively treated with no evidence of disease for > 5 years from enrollment.
4. Blood pressure that is not controlled despite > 2 oral agents (SBP >160 and DBP >90 documented during the screening period with no subsequent blood pressure readings >160/100).
5. History of seizure disorder or active use of anticonvulsants. Medications used to treat neuropathic pain such as gabapentin or pregabalin are allowed.
6. Serious inter-current infections or non-malignant medical illnesses that are uncontrolled.
7. Active psychiatric illness/social situations that would limit compliance with protocol requirements.
8. New York Heart Association (NYHA) class II, class III, or IV congestive heart failure (any symptomatic heart failure).
9. Concurrent therapy with strong inhibitors of Cytochrome P450 3A4 or CYP2C8 due to concerning possible drug-drug interactions.
10. Concurrent therapy with strong inducers of Cytochrome P450 3A4 due to concerning possible drug-drug interactions.
11. Presence of concurrent medical conditions requiring systemic glucocorticoids for immunosuppression (e.g. autoimmune diseases, organ transplantation) that is active and has required glucocorticoids in the last 6 months.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Response Rate of Subjects Receiving Relacorilant with Enzalutamide and Hormone Therapy | 24 weeks
  To determine if relacorilant (Rela) when added to androgen receptor signaling inhibition (ARSI) with enzalutamide (Enz) and androgen deprivation therapy (ADT) improves response rate compared to relacorilant with enzalutamide and ADT using both concurrent and historical controls. This outcome will be measured by assessing pathologic complete response rate (pCR) plus minimal residual disease (MRD) at radical prostatectomy (RP) after 24 weeks of neoadjuvant therapy.

SECONDARY OUTCOMES:
Radiographic Response Rate | 3 years and 9 months
  To determine if relacorliant when added to androgen receptor signaling inhibition (ARSI) improves radiographic and prostate-specific antigen (PSA) response rate compared to ARSI alone.
• To determine the 3-year biochemical recurrence-free survival (bRFS) and metastasis-free survival (MFS) rate with combination hormonal therapy with Rela + ARSI with Enz compared to ARSI with Enz alone | 3 years and 9 months
  To determine the 3-year biochemical recurrence-free survival (bRFS) and metastasis-free survival (MFS) rate with combination hormonal therapy with Rela + ARSI with Enz compared to ARSI with Enz alone.

CONTACTS AND LOCATIONS:
Overall Officials: Russell Szmulewitz, MD, Principal Investigator — University of Chicago
Locations (2):
- United States (2):
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF